CLINICAL TRIAL: NCT03632135
Title: Standard Chemotherapy Versus Chemotherapy Chosen by Cancer Stem Cell Chemosensitivity Testing in the Management of Patients With Recurrent Glioblastoma Multiforme (GBM).
Brief Title: Standard Chemotherapy vs. Chemotherapy Guided by Cancer Stem Cell Test in Recurrent Glioblastoma
Acronym: CSCRGBM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cordgenics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: CG01GBM
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Results first posted 2023-11-30 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Recurrent Glioblastoma
Keywords: ChemoID; Cancer stem cells; Drug response assay; Glioblastoma; Brain Cancer
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: parallel group randomized controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study investigators will be kept blind to the schedule. All participants will be screened by the ChemoID drug response assay; however, the treating physician will receive the ChemoID results only for those participants who are randomized to ChemoID-guided treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physician Choice treatment (Active Comparator): Participants will be treated with control chemotherapy treatment (standard-of-care chemotherapy chosen by the Physician from the provided list).
  Control chemotherapy treatment will be chosen from any of the following standard-of-care chemotherapy drugs or combinations:
  * Carboplatin;
  * Irinotecan;
  * Etoposide;
  * BCNU;
  * CCNU;
  * Temozolomide;
  * Procarbazine;
  * Vincristine;
  * Imatinib;
  * Procarbazine, CCNU, Vincristine;
  * Carboplatin, Irinotecan;
  * Carboplatin, Etoposide;
  * Temozolomide, Etoposide;
  * Temozolomide, Imatinib. The treating physician will NOT receive the ChemoID assay results from the ChemoID lab.
  Interventions: Diagnostic Test: ChemoID assay; Drug: Chemotherapy
- ChemoID-guided treatment (Experimental): Participants will be treated with ChemoID-guided standard-of-care chemotherapy drugs from the provided list.
  ChemoID-guided treatment will be chosen from the following standard-of-care chemotherapy drugs or combinations:
  * Carboplatin;
  * Irinotecan;
  * Etoposide;
  * BCNU;
  * CCNU;
  * Temozolomide;
  * Procarbazine;
  * Vincristine;
  * Imatinib;
  * Procarbazine, CCNU, Vincristine;
  * Carboplatin, Irinotecan;
  * Carboplatin, Etoposide;
  * Temozolomide, Etoposide;
  * Temozolomide, Imatinib.
  The treating physician will receive the ChemoID assay results from the ChemoID lab.
  Interventions: Diagnostic Test: ChemoID assay; Drug: Chemotherapy

INTERVENTIONS:
Diagnostic Test: ChemoID assay — The ChemoID test is a CLIA-certified and CAP-accredited drug response assay performed by a hospital clinical pathology laboratory that uses a patient's live tumor cells to indicate which chemotherapy agent (or combinations) will kill not only bulk of tumor cells, but importantly the cancer stem cells (CSCs) that are known to cause cancer to recur. During the assay, cancer stem cells and bulk tumor cells from an individual patient are exposed to FDA-approved chemotherapy drugs.
  The test measures the cytotoxic effect of actual doses of standard-of-care chemotherapies. The ChemoID drug response assay reports a prioritized list of effective and ineffective chemotherapies. The test is designed to target cancer stem cells to mitigate tumor relapse.
Drug: Chemotherapy — Chemotherapies chosen by Physician or ChemoID assay are in the same list of FDA approved drugs to treat recurrent high-grade glioma
  Other Names: Cytotoxic chemotherapy drugs

SUMMARY:
The purpose of this clinical study is to confirm the utility of chemosensitivity tumor testing on cancer stem cells (ChemoID) as a predictor of clinical response in poor prognosis malignant brain tumors such as recurrent glioblastoma (GBM).

DETAILED DESCRIPTION:
This study is designed as a parallel group randomized controlled clinical trial to determine if recurrent Glioblastoma (GBM) patients treated with drugs predicted by the ChemoID assay will have better outcomes than patients treated with standard-of-care control therapy chosen by the Physician.

Upon obtaining informed consent, all eligible participants affected by recurrent GBM will have a tumor biopsy to undergo ChemoID drug response testing with multiple FDA-approved chemotherapeutic agents.

Eligible participants will be randomized to a standard treatment arm with control treatment (chemotherapy chosen by the Physician from a provided list), or to a study arm of FDA-approved drugs selected by the ChemoID drug response assay.

ELIGIBILITY:
Inclusion Criteria:

1. Men and Women and members of all ethnic groups who are at least 18 years old at the time of enrollment are eligible for this trial;
2. Informed consent obtained and signed;
3. Willing and able to commit to study procedures including long-term follow-up visit(s);
4. Histopathologically confirmed 2016-WHO grade III recurrent glioma, and grade IV recurrent glioblastoma (GBM), inclusive of Gliosarcoma
5. In all cases, the diagnosis must be confirmed by a pathologist.
6. Recurrent surgically resectable tumor and/or biopsy;
7. Participants who have undergone surgical resection should have received an MRI or a scan after surgery in order to visualize residual tumor. If not, the operative report must be available;
8. Prior to surgery there was imaging evidence of measurable progressive disease (PD);
9. Start of radiotherapy, if indicated, must occur at least 2 weeks after surgery and/or biopsy;
10. Estimated survival of at least 3 months;
11. Hgb > 9 gm; absolute neutrophil count (ANC) > 1500/μl; platelets > 100,000; Creatinine < 1.5 times the upper limit of laboratory normal value; Bilirubin < 2 times the upper limit of laboratory normal value; serum glutamate pyruvate transaminase (SGPT) or serum glutamate oxaloacetate transaminase (SGOT) < 3 times the upper limit of laboratory normal value;
12. If indicated radiation therapy and chemotherapy must start within 8 weeks of tumor resection or biopsy.
13. Bevacizumab (Avastin) is allowed. If indicated it should be initiated at least 4 weeks post craniotomy or biopsy if the wound has healed well without any drainage or cellulitis;
14. The use of herbal preparation or tetrahydrocannabinol/cannabidiol is strongly discouraged, but not contraindicated;

Exclusion Criteria:

1. Subjects with newly diagnosed GBM
2. Pregnant women or nursing mothers cannot participate in the study. Women of childbearing age must have a negative pregnancy test within 72 hours prior to study entry. Women of childbearing potential must practice medically approved contraceptive precautions;
3. Abnormal hematological results at inclusion with: Neutrophils < 1,500/mm3; Blood-platelets < 100,000/mm3
4. Severe or chronic renal insufficiency (creatinine clearance ≤ 30 ml/min);
5. Patient unable to follow procedures, visits, examinations described in the study;
6. Any usual formal indication against imaging examinations (important claustrophobia, pacemaker);
7. History of another malignancy in the previous 2 years, with a disease-free interval of < 2 years. Patients with prior history of in situ cancer or basal or squamous cell skin cancer, any time prior to screening, are eligible;
8. OPTUNE device is not permitted in the study;
9. Patients cannot participate to any clinical trials utilizing a liquid biomarker or imaging studies that impact the overall survival.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tulika Ranjan, MD, Principal Investigator — Allegheny Health Network
Locations (13):
- United States (13):
  - Kaiser Permanente, Los Angeles, California
  - Keck School of Medicine of the University of Southern California, Los Angeles, California
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - Maine Medical Center Research Institute, Scarborough, Maine
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - Toledo University, Toledo, Ohio
  - Providence Cancer Center Oncology, Portland, Oregon
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - The Penn State Univeristy College of Medicine, Hershey, Pennsylvania
  - Thomas Jefferson University Hospitals, Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Charleston Area Medical Center, Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Howard CM, Valluri J, Alberico A, Julien T, Mazagri R, Marsh R, Alastair H, Cortese A, Griswold M, Wang W, Denning K, Brown L, Claudio PP. Analysis of Chemopredictive Assay for Targeting Cancer Stem Cells in Glioblastoma Patients. Transl Oncol. 2017 Apr;10(2):241-254. doi: 10.1016/j.tranon.2017.01.008. Epub 2017 Feb 12. PMID 28199863
- [Background] Ranjan T, Howard CM, Yu A, Xu L, Aziz K, Jho D, Leonardo J, Hameed MA, Karlovits SM, Wegner RE, Fuhrer R, Lirette ST, Denning KL, Valluri J, Claudio PP. Cancer Stem Cell Chemotherapeutics Assay for Prospective Treatment of Recurrent Glioblastoma and Progressive Anaplastic Glioma: A Single-Institution Case Series. Transl Oncol. 2020 Apr;13(4):100755. doi: 10.1016/j.tranon.2020.100755. Epub 2020 Mar 17. PMID 32197147
- [Background] Ranjan T, Yu A, Elhamdani S, Howard CM, Lirette ST, Denning KL, Valluri J, Claudio PP. Treatment of unmethylated MGMT-promoter recurrent glioblastoma with cancer stem cell assay-guided chemotherapy and the impact on patients' healthcare costs. Neurooncol Adv. 2023 May 12;5(1):vdad055. doi: 10.1093/noajnl/vdad055. eCollection 2023 Jan-Dec. PMID 37287692
- [Result] Ranjan T, Sengupta S, Glantz MJ, Green RM, Yu A, Aregawi D, Chaudhary R, Chen R, Zuccarello M, Lu-Emerson C, Moulding HD, Belman N, Glass J, Mammoser A, Anderson M, Valluri J, Marko N, Schroeder J, Jubelirer S, Chow F, Claudio PP, Alberico AM, Lirette ST, Denning KL, Howard CM. Cancer stem cell assay-guided chemotherapy improves survival of patients with recurrent glioblastoma in a randomized trial. Cell Rep Med. 2023 May 16;4(5):101025. doi: 10.1016/j.xcrm.2023.101025. Epub 2023 May 2. PMID 37137304

RESULTS

PARTICIPANT FLOW:
Groups:
- Physician Choice Treatment: Participants will be treated with control chemotherapy treatment (standard-of-care chemotherapy chosen by the Physician from the provided list).
  * Carboplatin;
  * Irinotecan;
  * Etoposide;
  * BCNU;
  * CCNU;
  * Temozolomide;
  * Procarbazine;
  * Vincristine;
  * Imatinib;
  * Procarbazine, CCNU, Vincristine;
  * Carboplatin, Irinotecan;
  * Carboplatin, Etoposide;
  * Temozolomide, Etoposide;
  * Temozolomide, Imatinib. The treating physician will NOT receive the ChemoID assay results from the ChemoID lab.
  ChemoID assay: The ChemoID test is a CLIA-certified and CAP-accredited drug response assay performed by a hospital clinical pathology laboratory that uses patient's live tumor cells to indicate which chemotherapy agent (or combinations) will kill not only bulk of tumor cells, but importantly the cancer stem cells (CSCs) that are known to cause cancer to recur. During the assay, cancer stem cells and bulk tumor cells from an individual patient are exposed to FDA-approved chemotherapy drugs.
  The test measures the cytotoxic effect of actual doses of standard-of-care chemotherapies. The ChemoID drug response assay reports a prioritized list of effective and ineffective chemotherapies. The test is designed to target cancer stem cells to mitigate tumor relapse.
  Chemotherapy: Chemotherapies chosen by Physician or ChemoID assay are in the same list of FDA approved drugs to treat recurrent GBM
- ChemoID-guided Treatment: Participants will be treated with ChemoID-guided standard-of-care chemotherapy drugs from the provided list.
  * Carboplatin;
  * Irinotecan;
  * Etoposide;
  * BCNU;
  * CCNU;
  * Temozolomide;
  * Procarbazine;
  * Vincristine;
  * Imatinib;
  * Procarbazine, CCNU, Vincristine;
  * Carboplatin, Irinotecan;
  * Carboplatin, Etoposide;
  * Temozolomide, Etoposide;
  * Temozolomide, Imatinib.
  The treating physician will receive the ChemoID assay results from the ChemoID lab.
  ChemoID assay: The ChemoID test is a CLIA-certified and CAP-accredited drug response assay performed by a hospital clinical pathology laboratory that uses patient's live tumor cells to indicate which chemotherapy agent (or combinations) will kill not only bulk of tumor cells, but importantly the cancer stem cells (CSCs) that are known to cause cancer to recur. During the assay, cancer stem cells and bulk tumor cells from an individual patient are exposed to FDA-approved chemotherapy drugs.
  The test measures the cytotoxic effect of actual doses of standard-of-care chemotherapies. The ChemoID drug response assay reports a prioritized list of effective and ineffective chemotherapies. The test is designed to target cancer stem cells to mitigate tumor relapse.
  Chemotherapy: Chemotherapies chosen by Physician or ChemoID assay are in the same list of FDA approved drugs to treat recurrent GBM
Period: Overall Study
Arm/Group | Physician Choice Treatment | ChemoID-guided Treatment
Started | 35 | 43
Completed | 35 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: subjects affected by recurrent GBM
Groups:
- Physician Choice Treatment: Participants will be treated with standard-of-care chemotherapy chosen by the Physician from the provided list.
  * Carboplatin;
  * Irinotecan;
  * Etoposide;
  * BCNU;
  * CCNU;
  * Temozolomide;
  * Procarbazine;
  * Vincristine;
  * Imatinib;
  * Procarbazine, CCNU, Vincristine;
  * Carboplatin, Irinotecan;
  * Carboplatin, Etoposide;
  * Temozolomide, Etoposide;
  * Temozolomide, Imatinib. The treating physician will NOT receive the ChemoID assay results from the ChemoID lab.
  ChemoID assay: The ChemoID test is a CLIA-certified and CAP-accredited drug response assay performed by a hospital clinical pathology laboratory that uses patient's live tumor cells to indicate which chemotherapy agent (or combinations) will kill not only bulk of tumor cells, but importantly the cancer stem cells (CSCs) that are known to cause cancer to recur. During the assay, cancer stem cells and bulk tumor cells from an individual patient are exposed to FDA-approved chemotherapy drugs.
  The test measures the cytotoxic effect of actual doses of standard-of-care chemotherapies. The ChemoID drug response assay reports a prioritized list of effective and ineffective chemotherapies. The test is designed to target cancer stem cells to mitigate tumor relapse.
  Chemotherapy: Chemotherapies chosen by Physician or ChemoID assay are in the same list of FDA approved drugs to treat recurrent Glioblastoma
- ChemoID-guided Treatment: Participants will be treated with ChemoID-guided standard-of-care chemotherapy drugs from the provided list.
  * Carboplatin;
  * Irinotecan;
  * Etoposide;
  * BCNU;
  * CCNU;
  * Temozolomide;
  * Procarbazine;
  * Vincristine;
  * Imatinib;
  * Procarbazine, CCNU, Vincristine;
  * Carboplatin, Irinotecan;
  * Carboplatin, Etoposide;
  * Temozolomide, Etoposide;
  * Temozolomide, Imatinib.
  The treating physician will receive the ChemoID assay results from the ChemoID lab.
  ChemoID assay: The ChemoID test is a CLIA-certified and CAP-accredited drug response assay performed by a hospital clinical pathology laboratory that uses patient's live tumor cells to indicate which chemotherapy agent (or combinations) will kill not only bulk of tumor cells, but importantly the cancer stem cells (CSCs) that are known to cause cancer to recur. During the assay, cancer stem cells and bulk tumor cells from an individual patient are exposed to FDA-approved chemotherapy drugs.
  The test measures the cytotoxic effect of actual doses of standard-of-care chemotherapies. The ChemoID drug response assay reports a prioritized list of effective and ineffective chemotherapies. The test is designed to target cancer stem cells to mitigate tumor relapse.
  Chemotherapy: Chemotherapies chosen by Physician or ChemoID assay are in the same list of FDA approved drugs to treat recurrent Glioblastoma
- Total: Total of all reporting groups
Arm/Group | Physician Choice Treatment | ChemoID-guided Treatment | Total
Number analyzed (Participants) | 35 | 43 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 5 | 15
  >=65 years | 25 | 38 | 63
Age, Continuous [Median (Standard Deviation); unit: years] | 55 (11) | 61 (13) | 59 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 21 | 28 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
  Black or African American | 1 | 0 | 1
  White | 31 | 36 | 67
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 43 | 78

OUTCOME MEASURES:

1. Primary Outcome: Median Overall Survival (OS)
Description: Overall survival (OS) in recurrent GBM patients who have had a ChemoID assay-guided treatment compared to standard therapy chosen by the physician.
Time Frame: 36 months
Population: Predetermined interim analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Physician Choice Treatment | ChemoID-guided Treatment
Number analyzed (Participants) | 35 | 43
months | 7.5 [3.5 to 11.5] | 12 [10.8 to 13.2]

2. Secondary Outcome: Median Progression Free Survival (PFS)
Description: Median Progression Free Survival in recurrent GBM patients who have had a ChemoID assay-guided treatment compared to standard therapy chosen by the physician.
Time Frame: 36 months
Population: final analysis
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Physician Choice Treatment: Participants will be treated with control chemotherapy treatment (standard-of-care chemotherapy chosen by the Physician from the provided list).
  Control chemotherapy treatment will be chosen from any of the following standard-of-care chemotherapy drugs or combinations:
  * Carboplatin;
  * Irinotecan;
  * Etoposide;
  * BCNU;
  * CCNU;
  * Temozolomide;
  * Procarbazine;
  * Vincristine;
  * Imatinib;
  * Procarbazine, CCNU, Vincristine;
  * Carboplatin, Irinotecan;
  * Carboplatin, Etoposide;
  * Temozolomide, Etoposide;
  * Temozolomide, Imatinib.
  The treating physician will NOT receive the ChemoID assay results from the ChemoID lab.
  ChemoID assay: The ChemoID test is a CLIA-certified and CAP-accredited drug response assay performed by a hospital clinical pathology laboratory that uses a patient's live tumor cells to indicate which chemotherapy agent (or combinations) will kill not only bulk of tumor cells, but importantly the cancer stem cells (CSCs) that are known to cause cancer to recur. During the assay, cancer stem cells and bulk tumor cells from an individual patient are exposed to FDA-approved chemotherapy drugs.
  The test measures the cytotoxic effect of actual doses of standard-of-care chemotherapies. The ChemoID drug response assay reports a prioritized list of effective and ineffective chemotherapies. The test is designed to target cancer stem cells to mitigate tumor relapse.
- ChemoID-guided Treatment: Participants will be treated with ChemoID-guided standard-of-care chemotherapy drugs from the provided list.
  ChemoID-guided treatment will be chosen from the following standard-of-care chemotherapy drugs or combinations:
  * Carboplatin;
  * Irinotecan;
  * Etoposide;
  * BCNU;
  * CCNU;
  * Temozolomide;
  * Procarbazine;
  * Vincristine;
  * Imatinib;
  * Procarbazine, CCNU, Vincristine;
  * Carboplatin, Irinotecan;
  * Carboplatin, Etoposide;
  * Temozolomide, Etoposide;
  * Temozolomide, Imatinib.
  The treating physician will receive the ChemoID assay results from the ChemoID lab.
  ChemoID assay: The ChemoID test is a CLIA-certified and CAP-accredited drug response assay performed by a hospital clinical pathology laboratory that uses a patient's live tumor cells to indicate which chemotherapy agent (or combinations) will kill not only bulk of tumor cells, but importantly the cancer stem cells (CSCs) that are known to cause cancer to recur. During the assay, cancer stem cells and bulk tumor cells from an individual patient are exposed to FDA-approved chemotherapy drugs.
  The test measures the cytotoxic effect of actual doses of standard-of-care chemotherapies. The ChemoID drug response assay reports a prioritized list of effective and ineffective chemotherapies. The test is designed to target cancer stem cells to mitigate tumor relapse.
Arm/Group | Physician Choice Treatment | ChemoID-guided Treatment
Number analyzed (Participants) | 35 | 43
months | 3.5 [1.9 to 5.1] | 10.1 [4.8 to 15.4]

ADVERSE EVENTS:
Time Frame: 5 years
Description: Clinical adverse events due to standard-of-care drugs (AEs) was monitored throughout the study. This study utilized the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 for CTEP-AERS (CTEP Adverse Event Reporting System) CAERs reporting of adverse events (AEs), located on the CTEP web site, http://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm. All appropriate treatment areas should have access to a copy of the CTCAE version 5.0.
Groups:
- Physician Choice Treatment: Participants will be treated with control chemotherapy treatment (standard-of-care chemotherapy chosen by the Physician from the provided list).
  * Carboplatin;
  * Irinotecan;
  * Etoposide;
  * BCNU;
  * CCNU;
  * Temozolomide;
  * Procarbazine;
  * Vincristine;
  * Imatinib;
  * Procarbazine, CCNU, Vincristine;
  * Carboplatin, Irinotecan;
  * Carboplatin, Etoposide;
  * Temozolomide, Etoposide;
  * Temozolomide, Imatinib. The treating physician will NOT receive the ChemoID assay results from the ChemoID lab.
  ChemoID assay: The ChemoID test is a CLIA-certified and CAP-accredited drug response assay performed by a hospital clinical pathology laboratory that uses patient's live tumor cells to indicate which chemotherapy agent (or combinations) will kill not only bulk of tumor cells, but importantly the cancer stem cells (CSCs) that are known to cause cancer to recur. During the assay, cancer stem cells and bulk tumor cells from an individual patient are exposed to FDA-approved chemotherapy drugs.
  The test measures the cytotoxic effect of actual doses of standard-of-care chemotherapies. The ChemoID drug response assay reports a prioritized list of effective and ineffective chemotherapies. The test is designed to target cancer stem cells to mitigate tumor relapse.
  Chemotherapy: Chemotherapies chosen by Physician or ChemoID assay are in the same list of FDA approved drugs to treat recurrent glioblastoma
Arm/Group | Physician Choice Treatment | ChemoID-guided Treatment
All-Cause Mortality (participants affected / at risk) | 35/35 | 43/43
Serious Adverse Events (participants affected / at risk) | 12/35 | 18/43
Other Adverse Events (participants affected / at risk) | 6/35 | 5/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physician Choice Treatment (N=35) | ChemoID-guided Treatment (N=43)
Low White blood cell count (Blood and lymphatic system disorders) | 8 (22) | 9 (12)
Low platelet count (Blood and lymphatic system disorders) | 7 (7) | 4 (5)
ALT increased (Hepatobiliary disorders) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Thromboembolia (Vascular disorders) | 0 (0) | 1 (1)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physician Choice Treatment (N=35) | ChemoID-guided Treatment (N=43)
Low white blood cells count (Blood and lymphatic system disorders) | 3 (5) | 2 (3)
Fatigue (General disorders) | 3 (4) | 1 (1)
Nausea (General disorders) | 1 (2) | 1 (1)
Decreased hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 2 (4) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (2) | 2 (2)
Neuropathy (Nervous system disorders) | 2 (2) | 2 (2)
Anorexia (General disorders) | 1 (1) | 1 (1)
weight loss (General disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 1 (2) | 1 (1)
Hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
weakness (General disorders) | 1 (2) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-01-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT03632135/Prot_SAP_ICF_001.pdf